CLINICAL TRIAL: NCT04392362
Title: A Randomised Controlled Trial of the Standard Versus a Simplified Adenosine Administration Method in the Treatment of Adult Patients With Supra- Ventricular Tachycardia (SVT)
Brief Title: A Trial to Compare American Heart Association (AHA) and Simple (SIM)Method to Give Adenosine to Treat Supra-ventricular Tachycardia (SVT)
Acronym: AHAvsSIM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pretoria (Other)
Responsible Party: Principal Investigator, Amanda Makhubela, MD, Principal investigator, University of Pretoria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPretoria
Record Dates: First submitted 2020-04-21; First posted 2020-05-18 (Actual); Results first posted 2021-06-25 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Supra-ventricular Tachycardia
MeSH Terms: interventions — Adenosine

STUDY DESIGN:
Intervention Model Description: Randomizes Control trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Method of giving adenosine at 6mg then 12mg repeated twice to abort svt Intervention is giving the drug in a simplified method mixing it with 20 ml saline as a whole flush
  Interventions: Drug: Adenosine
- Control group (Active Comparator): Giving adenosine Ising the recommended AHA two syringe method
  Interventions: Drug: Adenosine

INTERVENTIONS:
Drug: Adenosine — A vial of adenosine with 6mg

SUMMARY:
Study to compare non inferiority of giving adenosine with the simplified method vs the AHA method

DETAILED DESCRIPTION:
tle: A randomised controlled trial of the standard versus a simplified adenosine administration method in the treatment of adult patients with supra- ventricular tachycardia (SVT

ELIGIBILITY:
Inclusion Criteria:

* Svt
* normal blood pressure
* normal mentation
* Give consent

Exclusion Criteria:

* recent coffee
* Allergy to adenosine
* Asthma
* cardiac operations

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-12-16 (Actual); Study Completion 2020-12-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Steve Biko hospital, Pretoria, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neumar RW, Otto CW, Link MS, Kronick SL, Shuster M, Callaway CW, Kudenchuk PJ, Ornato JP, McNally B, Silvers SM, Passman RS, White RD, Hess EP, Tang W, Davis D, Sinz E, Morrison LJ. Part 8: adult advanced cardiovascular life support: 2010 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2010 Nov 2;122(18 Suppl 3):S729-67. doi: 10.1161/CIRCULATIONAHA.110.970988. PMID 20956224
- [Background] McDowell M, Mokszycki R, Greenberg A, Hormese M, Lomotan N, Lyons N. Single-syringe Administration of Diluted Adenosine. Acad Emerg Med. 2020 Jan;27(1):61-63. doi: 10.1111/acem.13879. Epub 2019 Nov 25. No abstract available. PMID 31665806
- [Background] Page RL, Joglar JA, Caldwell MA, Calkins H, Conti JB, Deal BJ, Estes NA 3rd, Field ME, Goldberger ZD, Hammill SC, Indik JH, Lindsay BD, Olshansky B, Russo AM, Shen WK, Tracy CM, Al-Khatib SM; Evidence Review Committee Chairdouble dagger. 2015 ACC/AHA/HRS Guideline for the Management of Adult Patients With Supraventricular Tachycardia: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Rhythm Society. Circulation. 2016 Apr 5;133(14):e506-74. doi: 10.1161/CIR.0000000000000311. Epub 2015 Sep 23. No abstract available. PMID 26399663
- [Background] Kaltenbach M, Hutchinson DJ, Bollinger JE, Zhao F. Stability of diluted adenosine solutions in polyvinyl chloride infusion bags. Am J Health Syst Pharm. 2011 Aug 15;68(16):1533-6. doi: 10.2146/ajhp100573. PMID 21817085
- [Background] Ketkar VA, Kolling WM, Nardviriyakul N, VanDer Kamp K, Wurster DE. Stability of undiluted and diluted adenosine at three temperatures in syringes and bags. Am J Health Syst Pharm. 1998 Mar 1;55(5):466-70. doi: 10.1093/ajhp/55.5.466. PMID 9522931
- [Background] Appelboam A, Reuben A, Mann C, Gagg J, Ewings P, Barton A, Lobban T, Dayer M, Vickery J, Benger J; REVERT trial collaborators. Postural modification to the standard Valsalva manoeuvre for emergency treatment of supraventricular tachycardias (REVERT): a randomised controlled trial. Lancet. 2015 Oct 31;386(10005):1747-53. doi: 10.1016/S0140-6736(15)61485-4. Epub 2015 Aug 24. PMID 26314489
- [Background] Shaker H, Jahanian F, Fathi M, Zare M. Oral verapamil in paroxysmal supraventricular tachycardia recurrence control: a randomized clinical trial. Ther Adv Cardiovasc Dis. 2015 Feb;9(1):4-9. doi: 10.1177/1753944714553425. Epub 2014 Oct 8. PMID 25297337
- [Background] 10. Hayes B. Trick of the Trade: Combine Adenosine with the Flush. Available at: https://www.aliem.com/trick-of-trade-combine-adenosine-single-syringe/. Accessed March 7, 2020.
- [Background] 11. Weingart S. SVT: The New Hotness. Emcrit. 2015. Available at: https://emcrit.org/emcrit/new-hotnesses-for-svt/. Accessed March 7, 2020.
- [Background] Choi SC, Yoon SK, Kim GW, Hur JM, Baek KW, Jung YS. A convenient method of adenosine administration for paroxysmal supraventricular tachycardia. J Korean Soc Emerg Med. 2003; 14:224-7
- [Background] 5. American Heart Association. ACLS for Experienced Providers Manual and Resource Text. United States of America: 2013.
- [Result] Orejarena LA, Vidaillet H Jr, DeStefano F, Nordstrom DL, Vierkant RA, Smith PN, Hayes JJ. Paroxysmal supraventricular tachycardia in the general population. J Am Coll Cardiol. 1998 Jan;31(1):150-7. doi: 10.1016/s0735-1097(97)00422-1. PMID 9426034

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention/SIM Group: Giving adenosine 6mg premixed with saline flush to a total of 20ml and giving it as a rapid flush, then same method repeated twice with 12 mg adenosine if the SVT does not convert
  The group evaluated was the SIM or intervention group
- Control/AHA Group: Giving adenosine as 6mg in one syringe with a separate syringe with 20ml saline flush using a three way stop cock to connect the syringes. Adenosine is given first as a rapid push followed by another rapid flush from the saline. The same method to be repeated twice with 12 mg adenosine if the SVT does not convert after 10-15 seconds
  The group evaluated was the AHA or control group
Period: Overall Study
Arm/Group | Intervention/SIM Group | Control/AHA Group
Started | 23 | 7
Completed | 23 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Simplified Method: Method of giving adenosine at 6mg then 12mg repeated twice to abort svt Intervention is giving the drug in a simplified method mixing it with 20 ml saline as a whole flush
  Adenosine: A vial of adenosine with 6mg
- AHA Method: Giving adenosine Ising the recommended AHA two syringe method
  Adenosine: A vial of adenosine with 6mg
- Total: Total of all reporting groups
Arm/Group | Simplified Method | AHA Method | Total
Number analyzed (Participants) | 23 | 7 | 30
Age, Customized [Count of Participants; unit: Participants]
  18-59 years | 16 | 5 | 21
  60-80 years | 7 | 2 | 9
Sex: Female, Male [Count of Participants; unit: Participants] — Patients were male or female
  Participants
    Female | 18 | 5 | 23
    Male | 5 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants] — The races were African, Asian, Coloured
  Participants
    Race: American Indian or Alaska Native | 0 | 0 | 0
    Race: Asian | 9 | 2 | 11
    Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Race: Black or African American | 13 | 5 | 18
    Race: White | 0 | 0 | 0
    Race: More than one race | 1 | 0 | 1
    Race: Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Africa | 23 | 7 | 30

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients With First Dose Successful Termination of the Supraventricular Tachycardia to a Sinus Rhythm of Less Than 140 With the AHA Versus a Simplified Method of Adenosine Administration
Description: The primary outcome is the rhythm of conversion to a sinus rhythm less than 140 beat per minute.
Time Frame: 10 seconds
Measure: Number; unit: participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 23 | 7
participants | 13 | 4
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; The null hypothesis is that the AHA method is inferior to the SIM method but not lower than a pre calculated noninferiority delta of -0.12 (-12 %) and a 95% one sided confidence interval. Only 33 (instead of 151 for a power of 95%) patients could be enrolled with 25 in the SIM and 8 in the AHA arms, which resulted in an estimated power test of 59.08%; Test type: Non-Inferiority — The non-inferiority margin or delta was calculated as -0.12(-12%); p = 0.8982, Wilcoxon (Mann-Whitney) — 0.05 was the level of significance; Risk Ratio (RR) = 0.89

ADVERSE EVENTS:
Time Frame: 2 hours
Description: There were no major adverse events
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/7
Other Adverse Events (participants affected / at risk) | 23/23 | 7/7
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (N=23) | Control Group (N=7)
Feeling of impending doom, dizziness (Cardiac disorders) | 23 (23) | 7 (7) — Feeling of impending doom, dizziness

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/62/NCT04392362/Prot_SAP_000.pdf